CLINICAL TRIAL: NCT05674071
Title: Applying an Osteopathic Intervention to Improve Mild to Moderate Mental Health
Brief Title: Applying an Osteopathic Intervention to Improve Mental Health Symptoms: a Mixed-methods Feasibility Study Protocol.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swansea University (Other)
Collaborators: Osteopathic Foundation (Unknown); University College of Osteopathy (Other)
Responsible Party: Principal Investigator, Darren Edwards, Principle Investigator, Swansea University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DEdwardsOsteopathy
Record Dates: First submitted 2022-12-06; First posted 2023-01-06 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Mental Health Issue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Articulation/HVT (Experimental): This intervention will use articulation and high-velocity thrust techniques
  Interventions: Behavioral: Articulation/HVT
- Soft-tissue massage (Experimental): This intervention will use soft-tissue massage
  Interventions: Behavioral: Soft-tissue massage
- Craniosacral techniques (Experimental): This intervention will use craniosacral techniques
  Interventions: Behavioral: Craniosacral techniques
- Combination (Experimental): This intervention will use a combination of the three interventions: HVT, soft-tissue and craniosacral
  Interventions: Behavioral: Combination of the three interventions: HVT, soft-tissue and craniosacral techniques

INTERVENTIONS:
Behavioral: Articulation/HVT — Osteopathy 1
  Arms: Articulation/HVT
Behavioral: Soft-tissue massage — Osteopathy 2
  Arms: Soft-tissue massage
Behavioral: Craniosacral techniques — Osteopathy 3
  Arms: Craniosacral techniques
Behavioral: Combination of the three interventions: HVT, soft-tissue and craniosacral techniques — This intervention will use a combination of the three interventions: HVT, soft-tissue and craniosacral techniques
  Arms: Combination

SUMMARY:
Applying an osteopathic intervention to improve mild to moderate mental health symptoms: a mixed-methods feasibility study protocol.

DETAILED DESCRIPTION:
Introduction: Mental health services are stretched in the UK and in need of support. One approach that could improve mental health symptoms is osteopathy. Research suggests that osteopathy influences psychophysiological factors, which could lead to improvements in mental health. The first objective of this protocol is to investigate the feasibility and acceptability of four osteopathic interventions. A secondary aim is to evaluate the interventions' effectiveness in improving psychophysiological and mental health outcomes.

Methods and analysis: This study will be an explanatory mixed-methods design. Participants will be 30 adults who have mild to moderate mental health symptoms and not experiencing any issues with pain. The feasibility and acceptability of the interventions will be the first primary outcome. Secondary outcomes will be physiological measures including heart rate variability (HRV), interoceptive accuracy (IAc) and blood pressure (BP). Psychological outcomes will also be measured by standardised questionnaires. These are being collected pre-and post-intervention. Additional outcomes will include recruitment rates and any adverse events that occur during the study. Participants will be randomised to one of four interventions. These are: high-velocity and articulation techniques (HVAT), soft-tissue massage (STM), craniosacral therapy (CST), and a combination of these three approaches. Participants will be interviewed about their experiences of the study and interventions to aid in assessing the feasibility and acceptability.

Discussion: This study will assess the feasibility and acceptability of conducting osteopathic interventions for improving mental health outcomes. These results from this will help to inform the running of a future randomised controlled trial. The study will also be producing original data which could provide preliminary evidence whether osteopathic approaches are of benefit to individual's mental health, even if they are pain-free.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate mental health symptoms as measured by DASS
* Ability to read/write English.

Exclusion Criteria:

* No mental health symptoms or severe mental health symptoms (as measured by DASS)
* acute or chronic pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of study recruitment | 3 months
  Recruitment rate
Feasibility of time to complete study | 3 months
  Time to complete questionnaires
Feasibility of study data collection | 3 months
  Missing data reported
Feasibility of assessing physiological measurements | 3 months
  Time to take physiological measurements
Acceptability of intervention to participants | 3 months
  Feedback from participants in qualitative interviews
Acceptability of intervention and risk factors | 3 months
  Adverse events reported

SECONDARY OUTCOMES:
Depression Anxiety and Stress Scale (DASS) | 3 months
  Measure of depression, anxiety and stress. Scores range from 0-21 for each of the 3 sub scales and higher scores indicate greater levels of depression, anxiety or stress.
Positive and negative affect schedule (PANAS) | 3 months
  Measure of positive and negative affect. Scores range from 10-50 for each of the 2 sub scales and higher scores indicate higher levels of positive and negative affect.
Acceptance and action questionnaire (AAQ) | 3 months
  Measure of psychological inflexibility. Scores range from 7-49 and higher scores indicate higher levels of psychological inflexibility.
Self as context scale (SACS) | 3 months
  Measure of self-as-context and perspective taking. Has two sub scales of centering and transcending ranging from 5-35, with higher scores indicating greater levels of these.
Multidimensional Assessment of Interoceptive Awareness (MAIA) | 3 months
  Measure of interoceptive awareness. Uses 8 sub scales and higher scores indicate greater levels of each domain of interoceptive awareness.
Heart rate variability | 3 months
  Measure by time-domain: root mean square of successive interval differences (RMSSD) and frequency domain: low frequency to high frequency ratio.
Interoceptive accuracy | 3 months
  Measured using heartbeat detection task
Blood pressure | 3 months
  Participants blood pressure will be recorded according to NICE guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Darren Edwards, PhD, Principal Investigator — Swansea University
Locations (1):
- Swansea University, Swansea, Select State, United Kingdom

REFERENCES:
- [Derived] Hope-Bell J, Draper-Rodi J, Edwards DJ. Applying an osteopathic intervention to improve mild to moderate mental health symptoms: a mixed-methods feasibility randomised trial. Chiropr Man Therap. 2024 Nov 6;32(1):32. doi: 10.1186/s12998-024-00556-x. PMID 39506737
- [Derived] Hope-Bell J, Draper-Rodi J, Edwards DJ. Applying an osteopathic intervention to improve mild to moderate mental health symptoms: a mixed-methods feasibility study protocol. BMJ Open. 2023 Jun 27;13(6):e071680. doi: 10.1136/bmjopen-2023-071680. PMID 37369421